CLINICAL TRIAL: NCT06538467
Title: Comparison of Architectural and Performance Adaptations of Hip Extension Exercise Under Gravitational or Inertial Loading Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rodrigo Martín-San-Agustin, Assistant Professor of Physiotherapy, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H1551979435533
Record Dates: First submitted 2024-07-27; First posted 2024-08-05 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Injury;Sports
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inertial (Experimental): Hip extension exercise performed under inertial loading conditions using the EPTE Inertial Concept (Ionclinics SL, L'Alcudia, Spain) during six weeks with two sessions per week. The EPTE Inertial Concept is an inertial device that combines a series of output pulleys and telescopic arms, capable of implementing 6 disks of different weights and radii.
  Interventions: Other: Hip extension exercise with inertial load
- Gravitational (Experimental): Hip extension exercise performed under gravitational loading conditions using free-weight equipment during six weeks with two sessions per week.
  Interventions: Other: Hip extension exercise with gravitational load
- Control (No Intervention): Participans was advised to continue their regular levels of physical activity but not to perform any lower body resistance training

INTERVENTIONS:
Other: Hip extension exercise with inertial load — Hip extension exercise with inertial load
  Arms: Inertial
Other: Hip extension exercise with gravitational load — Hip extension exercise with gravitational load
  Arms: Gravitational

SUMMARY:
The main objective of this study is to investigate training-induced adaptations in Biceps femoris long head (BFlh) architecture and performance measures such as muscle strength, jumping, and power variables after following 6 weeks of resistance training program with gravitational or inertial hip extension (HE) exercise and a subsequent detraining period, comparing those adaptations with a control group. In addition, this study aims to determine the time course of BFlh architectural adaptations throughout a 6-week training intervention.

ELIGIBILITY:
Inclusion Criteria:

* at least two years of resistance training experience
* not have any injury, disease or pain that could reduce their maximal effort

Exclusion Criteria:

* history of injury to the lower limbs (including the hamstrings), wrist, or back in the past 18 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Fascicle length | Baseline, at weeks 2 and 3 of the intervention, at the end of the 6 weeks of training and 4 weeks after this (detraining period)
  Two-dimensional images of the Biceps femoris long head (BFlh) architecture were captured using B-mode ultrasonography. All imaging was conducted with participants lying prone with their hips and knees in a neutral and fully extended position.Three ultrasound images were taken and stored for analysis through the ImageJ software (National Institutes of Health, USA).
  The most visible fascicle in each image was used for measurement of fascicle pennation angle (i.e., angle between the fascicle and the intermediate aponeurosis) and estimation of fascicle length using a validated equation:
  FL = sin (AA + 90°) × MT ÷ sin (180° - (AA + 180° - PA))
Muscle Strength Assessment | Baseline, at the end of the 6 weeks of training and 4 weeks after this (detraining period)
  Knee flexion was assessed with subjects in prone position performing knee flexor maximal isometrics contractions with a knee angle of approximately 15 degrees. For hip extension, a resisted hip extension was requested with the subjects lying in the prone position with their legs straight. Hip adduction was evaluated in a supine position with the hips at 45º flexion, requesting an maximal isometrics contraction adduction with a resistance in the internal condyle.
Jump performance | Baseline, at the end of the 6 weeks of training and 4 weeks after this (detraining period)
  CMJ and SJ, utilizing the MyJump 2 application on an iPad Pro (at 240 frames per second, high-definition video resolution). In the CMJ, participants initiated the jump from a standing position, performed a preparatory movement by bending their knees to 90° flexion, and then jumped upward as high as possible without pausing between movements. Similarly, for the SJ, participants began from a standardized position with knees flexed at 90°, and then jumped as high as possible with hands on their hips. Throughout both tests, participants were instructed to maintain their hands on their hips to minimize lateral and horizontal displacement, ensuring accurate vertical jump measurement.
Power | Baseline, at the end of the 6 weeks of training and 4 weeks after this (detraining period)
  Power was calculated in both modalities (i.e., HE gravitational and inertial) as the product of velocity and force. The velocity was calculated using the MuscleLab 4020e linear encoder (Ergotest Technology AS, Porsgrunn, Norway). For gravitational loading (i.e. constant mass), the force was calculated as the product of mass and acceleration. For inertial loading, the force was calculated using a force gauge that was anchored along the rope, between a pulley and the proximal end of the second rope.
Soreness | From session 1 (the beginning of week 1) to session 12 (the end of week 6), at the beginning and end of each session.
  Participants were asked "How sore do you feel in your hamstrings?" and rated their soreness on a 10-point Likert Scale (1 = No Soreness, 3 = Minimal Soreness, 5 = Moderate Soreness, 8 = Very Sore, 10 = Extremely Sore)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Martín-San Agustín, Principal Investigator — University of Valencia
Locations (1):
- Rodrigo Martin-San Agustin, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No